CLINICAL TRIAL: NCT02491073
Title: Ex-vivo Study to Evaluate Serum Free Thyroxine (FT4) and Free Triiodothyronine (FT3) Measurements Using Equilibrium Dialysis (ED) and Automated Kit Assay for Subjects Treated With Eslicarbazeine Acetate
Brief Title: Study to Evaluate Serum Free Thyroxine (FT4) and Free Triiodothyronine (FT3) Measurements for Subjects Treated With Eslicarbazeine Acetate (ESL)
Status: Completed | Type: Observational
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEP093-451
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eslicarbazepine acetate treated
  Interventions: Other: blood draw
- Non-Eslicarbazepine acetate treated
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Investigate the possibility of assay artifacts impacting the measurement of thyroid hormones, in particular FT4 and FT3, in ESL treated subjects compared to non-ESL-treated subjects.

SUMMARY:
The purpose of this research study is to determine if the blood tests used to measure free thyroid hormone levels are affected by a drug called eslicarbazepine acetate. To determine if eslicarbazepine acetate interferes with these blood tests, blood samples will be analysed so that researchers can compare different types of lab tests that measure these thyroid hormones. Half of the people who participate in this study will already be taking eslicarbazepine acetate either as a study drug or as a prescription (Part 1) and the other half will be people who do not take eslicarbazepine acetate (Part 2).

DETAILED DESCRIPTION:
Part 1 of the study will enroll a minimum of 30 male and female subjects who have received at least 1200 mg once daily (QD) ESL over a minimum 6-week period (ESL-exposed subjects). Subjects, who meet study eligibility requirements and provide written consent, will provide blood samples for measurement of thyroid hormones, thyroxine binding globulins (TBG), serum pregnancy (female subjects of childbearing potential 1only), thyroid peroxidase (TPO) antibodies, and ESL metabolites (eslicarbazepine and (R)-licarbazepine).

Optional blood samples will be requested from subjects in Part 1 who provide genetic consent and are eligible to participate (as controls) in a separate rash registry protocol. These samples will be tested for HLA typing, genetic ancestry, and viral titers (including human herpes virus [HHV]-6, HHV-7, and Epstein-Barr virus [EBV]).

ESL metabolites will be determined by a validated liquid chromatography- tandem mass spectrometry (LC-MS/MS) assay. Levels of FT4 and FT3 in ESL-exposed serum will be assayed using the automated kit assay (Roche Cobas ECLIA kits FT4 II and FT3 III) and Equilibrium Dialysis (ED) method. FT4 and FT3 results measured by both methods will be compared to evaluate potential assay differences. Serum TSH, TT4, TT3, and TBG in ESL treated subject samples will also be measured using automated kit assays.

Part 2 of the study will enroll a minimum of 30 age (± 5 y) and gender-matched non-ESL exposed volunteers. Subjects, who meet study eligibility requirements and provide written consent, will provide a blood sample for measurement of thyroid hormones, TBG, serum pregnancy (female subjects of childbearing potential only), and TPO antibodies. Serum samples obtained from non-ESL exposed subjects will be split into 4 aliquots, one aliquot will be used as the control blank (unspiked) and the rest spiked with 3 levels (high, low, and a concentration representative of therapeutic levels also called middle) of eslicarbazepine (range approximately 5 to 18 μg/mL) and (R)-licarbazepine (range approximately 0.5 to 1.8 μg/mL). The low concentration for spiking the non-ESL exposed samples will be approximately 1 standard deviation (SD) below Cavg associated with the 800 mg dose in chronic use in the epilepsy population and the high concentration for spiking will be approximately 1 SD above Cavg associated with the 1200 mg dose.

After sample is spiked with eslicarbazepine and (R)-licarbazepine, serum FT4 and FT3 will be measured by the automated kit assay method, as well as ED method. FT4 and FT3 measured in non-spiked and spiked volunteer samples will be compared to detect potential in vitro artifacts. Serum TSH, TT4, TT3, and TBG in non-spiked and spiked volunteer samples will also be measured using automated kit assays.

ELIGIBILITY:
Inclusion Criteria:

* ESL-exposed Subjects

  1. Subject must give written informed consent and privacy authorization prior to participation in the study.
  2. Male or female patient (≥ 18 years of age) who has received at least 1200 mg QD ESL for at least 6 weeks and has not experienced any rash or other allergic reaction at the time of blood draw.
* Non-ESL-exposed Subjects

  1. Subject must give written informed consent and privacy authorization prior to participation in the study.
  2. Male or female healthy normal volunteer (≥ 18 years of age).

Exclusion Criteria:

* Both ESL-exposed and non-ESL exposed subjects

  1. Subject who does not tolerate venipuncture or Has poor venous access that would cause difficulty for collecting blood samples.
  2. Subject with a history of thyroid disease or clinical condition (eg, renal insufficiency, Sjogren's syndrome, lupus, rheumatoid arthritis, pernicious anemia etc.) that in the opinion of the Investigator may effect levels of thyroid hormones, TBG, and/or TPO antibodies.
  3. Female subject who is pregnant.
  4. Female subject with a positive urine pregnancy test at screening.
  5. Subject who received any excluded medication for at least 30 days prior to blood draw.
  6. Subject has experienced significant blood loss and/or donated blood within last 60 days of blood draw.
  7. Subject intends to donate blood or undergo elective surgery within next 30 days following blood draw.
  8. Subject has donated plasma within last 72 hours of blood draw or intends to donate plasma during study participation.
  9. Subject is, in the opinion of the Investigator, unsuitable in any other way to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and Females greater than or equal to 18 years of age, either exposed to drug or not exposed to drug
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (7):
- United States (7):
  - The More foundation/The Core Institute, Sun City, Arizona
  - Consultans in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - Mid-Atlantic Epilepsy Center, Bethesda, Maryland
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - CliniLabs, New York, New York
  - NeurologicalClinic of Texas, P.A., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Eslicarbazepine Acetate Exposed Subjects: Adult male and female subjects (greater than or equal to 18 years)who had received at least 1200 mg QD eslicarbazapine acetate (ESL) for at least 6 weeks and had not experienced any rash or other allergic reaction at the time of the blood draw
- Healthy Volunteers: Adult male and female healthy volunteer (greater than or equal to 18 years) not exposed to ESL at the time of blood draw
Period: Overall Study
Arm/Group | Eslicarbazepine Acetate Exposed Subjects | Healthy Volunteers
Started | 37 | 34
Completed | 36 | 34
Not Completed | 1 | 0
Not completed — screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: the analysis was done on the safety population group
Groups:
- Total: Total of all reporting groups
Arm/Group | Eslicarbazepine Acetate Treated | Non-Eslicarbazepine Acetate Treated | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.95) | 41.7 (14.64) | 41.8 (14.68)
Age, Customized [Number; unit: participants]
  <18 years of age | 0 | 0 | 0
  18-39 Years | 16 | 16 | 32
  40-65 Years | 13 | 13 | 26
  >65 Years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 20 | 23
  White | 26 | 6 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Concentrations of Free Thyroid Hormones (FT4 and FT3) as Measured by ED and Automated Kit Assay Method in ESL-exposed Subjects
Time Frame: 1 day
Population: Safety Population: The safety population consisted of all subjects who were enrolled in the study, did not test positive for serum pregnancy (female subjects of childbearing potential only) or TPO antibodies, and provided valid serum samples for evaluating the thyroid hormone assays
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Groups:
- Automated Kit Assay (AK) - ESL-exposed Subjects: Free thyroid hormone level in the serum sample of ESL-exposed subjects as measured by the automated kit assay
- Optimized Equilibrium Dialysis Method (ED)ESL-exposed Subjects: Free thyroid hormone level in the serum sample of ESL-exposed subjects as measured by the optimized equilibrium dialysis method
Arm/Group | Automated Kit Assay (AK) - ESL-exposed Subjects | Optimized Equilibrium Dialysis Method (ED)ESL-exposed Subjects
Number analyzed (Participants) | 31 | 31
pmol/L
  FT4: pmol/L | 12.29 (0.139) | 11.74 (0.244)
  FT3: pmol/L | 4.20 (0.112) | 3.65 (0.183)
Statistical Analysis 1: Comparison: Automated Kit Assay (AK) - ESL-exposed Subjects vs Optimized Equilibrium Dialysis Method (ED)ESL-exposed Subjects; There is no hypothesis testing in this study. The sample size was determined outside of statistical considerations; it was required by the U.S. Food and Drug Administration (FDA) in the New Drug Application 022416 Approval Letter issued on 08 November 2013 for PMR 2099-9; Test type: Other; p = 1.05, geometric mean ration; geometric mean ratio = 1.05, 90% CI 2-sided [0.98 to 1.09] — The parameter dispersion type:Geometric coefficient of variation Dispersion Value: FT4: 0.220; In each geometric mean ratio estimate, free thyroid hormone levels as measured by the automated kit assay represent the numerator; free thyroid hormone levels as measured by the optimized equilibrium dialysis method represent the denominator
Statistical Analysis 2: Comparison: Automated Kit Assay (AK) - ESL-exposed Subjects vs Optimized Equilibrium Dialysis Method (ED)ESL-exposed Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio; Geometric Mean Ratio = 1.15, 90% CI 2-sided [1.09 to 1.22] — parameter dispersion type: Geometric Coefficient of Variation Dispersion Value : FT3: 0.178; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Comparison of Concentrations of Free Thyroid Hormones (FT4 and FT3) as Measured by Automated Kit Assay in Non-ESL Exposed Subjects, With and Without the in Vitro Addition of Eslicarbazepine and (R)-Licarbazepine.
Time Frame: 1 day
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Groups:
- Non-spiked Serum(NS) Healthy Volunteers: Free thyroid hormone level in the serum sample of healthy volunteers which was not spiked with ESL metabolites
- Low-spiked Serum(LS)Healthy Volunteers: Free thyroid hormone level in the serum sample of healthy volunteers which was spiked with low level of ESL metabolites
- Mid-spiked Serum(MS)Healthy Volunteers: Free thyroid hormone level in the serum sample of healthy volunteers which was spiked with medium level of ESL metabolites
- High-spiked Serum(HS)Healthy Volunteers: Free thyroid hormone level in the serum sample of healthy volunteers which was spiked with high level of ESL metabolites
Arm/Group | Non-spiked Serum(NS) Healthy Volunteers | Low-spiked Serum(LS)Healthy Volunteers | Mid-spiked Serum(MS)Healthy Volunteers | High-spiked Serum(HS)Healthy Volunteers
Number analyzed (Participants) | 31 | 31 | 31 | 31
pmol/L
  FT4: pmo/L | 15.64 (0.146) | 15.84 (0.147) | 16.15 (0.146) | 16.49 (0.145)
  FT3: pmo/L | 4.92 (0.125) | 4.95 (0.128) | 5.00 (0.133) | 5.06 (0.122)
Statistical Analysis 1: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Low-spiked Serum(LS)Healthy Volunteers; FT4; Test type: Other — There is no hypothesis testing in this study. The sample size was determined outside of statistical considerations; it was required by the U.S. Food and Drug Administration (FDA) in the New Drug Application 022416 Approval Letter issued on 08 November 2013 for PMR 2099-9; Geometric Mean Ratio = 1.01, 90% CI 2-sided [1.01 to 1.03] — Parameter dispersion type: geometric coefficient of variation dispersion value 0.024; In each geometric mean ratio estimate, free thyroid hormone levels in the spiked serum samples (LS or MS or HS) represent the numerator; free thyroid hormone levels in non-spiked serum samples (NS) represent the denominator
Statistical Analysis 2: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; Geometric Mean Ratio = 1.03, 90% CI 2-sided [1.03 to 1.04] — parameter dispersion value - geometric coefficient of variation dispersion value - 0.020; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.05, 90% CI 2-sided [1.05 to 1.06] — parameter dispersion type - geometric coefficient variation dispersion value - 0.021; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Low-spiked Serum(LS)Healthy Volunteers; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [0.99 to 1.02] — parameter dispersion type -geometric coefficient of variation dispersion value - 0.040; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geotmetric mean ratio = 1.02, 90% CI 2-sided [1.00 to 1.03] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.041; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.03, 90% CI 2-sided [1.02 to 1.04] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.041; [other analysis details as in outcome 2, analysis 1]

3. Secondary Outcome: Comparison of Concentrations of TT4, and TT3 as Measured in Non-ESL-exposed Subject Samples, With or Without the in Vitro Addition of Eslicarbazepine and (R)-Licarbazepine.
Time Frame: 1 day
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmo/L
Groups:
- Non-spiked Serum(NS) Healthy Volunteers: thyroid hormone level in the serum sample of healthy volunteers which was not spiked with ESL metabolites
- Low-spiked Serum(LS)Healthy Volunteers: thyroid hormone level in the serum sample of healthy volunteers which was spiked with low level of ESL metabolites
- Mid-spiked Serum(MS)Healthy Volunteers: thyroid hormone level in the serum sample of healthy volunteers which was spiked with medium level of ESL metabolites
- High-spiked Serum(HS)Healthy Volunteers: thyroid hormone level in the serum sample of healthy volunteers which was spiked with high level of ESL metabolites
Arm/Group | Non-spiked Serum(NS) Healthy Volunteers | Low-spiked Serum(LS)Healthy Volunteers | Mid-spiked Serum(MS)Healthy Volunteers | High-spiked Serum(HS)Healthy Volunteers
Number analyzed (Participants) | 31 | 31 | 31 | 31
nmo/L
  TT4: nmo/L | 94.82 (0.177) | 95.10 (0.173) | 96.06 (0.169) | 94.82 (0.165)
  TT#: nmo/L | 1.69 (0.158) | 1.68 (0.158) | 1.68 (0.160) | 1.67 (0.161)
Statistical Analysis 1: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Low-spiked Serum(LS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value -0.018; In each geometric mean ratio estimate, thyroid hormone levels in the spiked serum samples (LS or MS or HS) represent the numerator; thyroid hormone levels in non-spiked serum samples (NS) represent the denominator
Statistical Analysis 2: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.018; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.018
Statistical Analysis 4: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Low-spiked Serum(LS)Healthy Volunteers; TT4; Test type: Other — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.00, 90% CI 2-sided [0.99 to 1.02] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.041; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; TT4; Test type: Other — [test comment as in outcome 2, analysis 1]; Slope = 1.01, 90% CI 2-sided [1.00 to 1.02] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.033; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; TT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [0.99 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.036; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Low-spiked Serum(LS)Healthy Volunteers; TT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 0.99, 90% CI 2-sided [0.98 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.047; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; TT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [0.98 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.043; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; TT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 0.99, 90% CI 2-sided [0.97 to 1.00] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.048; [other analysis details as in outcome 3, analysis 1]

4. Secondary Outcome: Comparison of Concentrations of Free Thyroid Hormones (FT4 and FT3) in Spiked and Unspiked Volunteer Samples Using ED and Automated Kit Assay.
Time Frame: 1 day
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Groups:
- Automated Kit Assay(AK)Non-spiked Serum(NS)Healthy Volunteers: Free thyroid hormone level as measured by the automated kit assay in the serum sample of healthy volunteers which was not spiked with ESL metabolites
- Optimized Equilibrium Dialysis Method(ED)(NS)Healthyvolunteer: Free thyroid hormone level as measured by the optimized equilibrium dialysis method in the serum sample of healthy volunteers which was not spiked with ESL metabolites
- Automated Kit Assay(AK)Low-spiked Serum(LS)Healthy Volunteers: Free thyroid hormone level as measured by the automated kit assay in the serum sample of healthy volunteers which was spiked with low level of ESL metabolites
- Optimized Equilibrium Dialysis Method(ED)(LS)Healthyvolunteer: Free thyroid hormone level as measured by the optimized equilibrium dialysis method in the serum sample of healthy volunteers which was spiked with low level of ESL metabolites
- Automated Kit Assay(AK)Med-spikedSerum(MS)Healthy Volunteers: Free thyroid hormone level as measured by the automated kit assay in the serum sample of healthy volunteers which was spiked with medium level of ESL metabolites
- Optimized Equilibrium Dialysis Method(ED)(MS)Healthyvolunteer: Free thyroid hormone level as measured by the optimized equilibrium dialysis method in the serum sample of healthy volunteers which was spiked with medium level of ESL metabolites
- Automated Kit Assay(AK)High-spikedSerum(HS)Healthy Volunteers: Free thyroid hormone level as measured by the automated kit assay in the serum sample of healthy volunteers which was spiked with high level of ESL metabolites
- Optimized Equilibrium Dialysis Method(ED)(HS)Healthyvolunteer: Free thyroid hormone level as measured by the optimized equilibrium dialysis method in the serum sample of healthy volunteers which was spiked with high level of ESL metabolites
Arm/Group | Automated Kit Assay(AK)Non-spiked Serum(NS)Healthy Volunteers | Optimized Equilibrium Dialysis Method(ED)(NS)Healthyvolunteer | Automated Kit Assay(AK)Low-spiked Serum(LS)Healthy Volunteers | Optimized Equilibrium Dialysis Method(ED)(LS)Healthyvolunteer | Automated Kit Assay(AK)Med-spikedSerum(MS)Healthy Volunteers | Optimized Equilibrium Dialysis Method(ED)(MS)Healthyvolunteer | Automated Kit Assay(AK)High-spikedSerum(HS)Healthy Volunteers | Optimized Equilibrium Dialysis Method(ED)(HS)Healthyvolunteer
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
pmol/L
  FT4 pmol/L | 15.64 (0.146) | 14.08 (0.193) | 15.84 (0.147) | 13.99 (0.204) | 16.15 (0.146) | 14.57 (0.254) | 16.49 (0.145) | 15.80 (0.232)
  FT3 pmol/L | 4.92 (0.125) | 4.06 (0.192) | 4.95 (0.128) | 3.47 (0.273) | 5.00 (0.133) | 4.20 (0.208) | 5.06 (0.122) | 4.27 (0.246)
Statistical Analysis 1: Comparison: Automated Kit Assay(AK)Non-spiked Serum(NS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(NS)Healthyvolunteer; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.11, 90% CI 2-sided [1.06 to 1.16] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.148; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Automated Kit Assay(AK)Low-spiked Serum(LS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(LS)Healthyvolunteer; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.13, 90% CI 2-sided [1.07 to 1.20] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.202; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Automated Kit Assay(AK)Med-spikedSerum(MS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(MS)Healthyvolunteer; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.11, 90% CI 2-sided [1.04 to 1.18] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.203; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Automated Kit Assay(AK)High-spikedSerum(HS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(HS)Healthyvolunteer; FT4; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.04, 90% CI 2-sided [0.99 to 1.10] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.179; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Automated Kit Assay(AK)Non-spiked Serum(NS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(NS)Healthyvolunteer; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.21, 90% CI 2-sided [1.15 to 1.52] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.178; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Automated Kit Assay(AK)Low-spiked Serum(LS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(LS)Healthyvolunteer; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.42, 90% CI 2-sided [1.33 to 1.52] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.224; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Automated Kit Assay(AK)Med-spikedSerum(MS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(MS)Healthyvolunteer; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.19, 90% CI 2-sided [1.12 to 1.27] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.203; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Automated Kit Assay(AK)High-spikedSerum(HS)Healthy Volunteers vs Optimized Equilibrium Dialysis Method(ED)(HS)Healthyvolunteer; FT3; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.19, 90% CI 2-sided [1.11 to 1.27] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.215; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Comparison of Concentrations of TSH,as Measured in Non-ESL-exposed Subject Samples, With or Without the in Vitro Addition of Eslicarbazepine and (R)-Licarbazepine.
Time Frame: 1 day
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mU/L
Arm/Group | Non-spiked Serum(NS) Healthy Volunteers | Low-spiked Serum(LS)Healthy Volunteers | Mid-spiked Serum(MS)Healthy Volunteers | High-spiked Serum(HS)Healthy Volunteers
Number analyzed (Participants) | 31 | 31 | 31 | 31
mU/L | 1.32 (0.566) | 1.33 (0.563) | 1.32 (0.569) | 1.33 (0.565)
Statistical Analysis 1: Comparison: Low-spiked Serum(LS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value -0.018; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs Mid-spiked Serum(MS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.018; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Non-spiked Serum(NS) Healthy Volunteers vs High-spiked Serum(HS)Healthy Volunteers; TSH; Test type: Other — [test comment as in outcome 2, analysis 1]; geometric mean ratio = 1.00, 90% CI 2-sided [1.00 to 1.01] — parameter dispersion type - geometric coefficient of variation dispersion value - 0.018

ADVERSE EVENTS:
Time Frame: One day
Description: Adverse events were collected on the same day as the study visit
Arm/Group | Eslicarbazepine Acetate Exposed Subjects | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34
Other Adverse Events (participants affected / at risk) | 1/37 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine Acetate Exposed Subjects (N=37) | Healthy Volunteers (N=34)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the study at all sites, institution and investigator shall be free to publish